CLINICAL TRIAL: NCT05755217
Title: Study of the Renal Physiological Response After Chocolate Consumption
Brief Title: Renal Ultrasound Response After Chocolate Consumption
Acronym: Choco
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gregoire Wuerzner; MD (Other)
Responsible Party: Sponsor-Investigator, Gregoire Wuerzner; MD, Professor Grégoire Wuerzner, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022-01359
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chocolate Consumption
Keywords: chronic kidney disease; doppler ultrasound; renal resistive index; handgrip test; dark chocolate; white chocolate; cocoa
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This study will be a single-blinded randomized cross-over study, comparing the renal physiological effects of dark chocolate (DC) with white chocolate (WC). Doppler ultrasounds will take place in the Service of Nephrology of the CHUV, between late morning and early afternoon. Healthy participants who meet the inclusion criteria will be divided in small groups of 3-4 persons according to the order of inclusion. CKD participants will be investigated separately. Every participant will sign an informed consent form before the beginning of the study
Who Masked: Investigator
Masking Description: The sonographer will be blinded for the study intervention (eg, dark or white chocolate consumption)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dark chocolate (Active Comparator): Single dose of 1g/kg of dark chocolate (70% cocoa, Lindt Excellence)
  Interventions: Dietary Supplement: Dark chocolate
- White chocolate (Placebo Comparator): Single dose of 1g/kg of white chocolate (4% cocoa, Nestle Galak).
  Interventions: Dietary Supplement: White chocolate

INTERVENTIONS:
Dietary Supplement: Dark chocolate — Single oral dose of 1g/kg of dark chocolate (70% cocoa).
  Arms: Dark chocolate
Dietary Supplement: White chocolate — Single oral dose of 1g/kg of white chocolate (4% cocoa).
  Arms: White chocolate

SUMMARY:
The consumption of dark chocolate (DC) has antihypertensive (3) and anti-inflammatory effects. Some studies also suggest that dark chocolate may also have cardiovascular benefits, but its physiological effects on the kidneys have not been studied in detail.

In this randomized, single-blinded, controlled, monocentric cross-over study we will investigate whether the ingestion of a single dose of dark chocolate (g/kg, max 70g) leads to alterations in renal perfusion and blood pressure two hours after its consumption in healthy volunteers and patients suffering from chronic kidney disease.

The Doppler-ultrasound assessed renal resistive index (RRI) will be used at baseline and two hours after chocolate consumption as an indirect measure of renal perfusion. Blood pressure and heart rate will be measured continuously using the Finapres® NOVA (Finapres Medical Systems, Enschede, The Netherlands) throughout the Doppler ultrasound examination.

In order to compare the effects of dark chocolate with those obtained with white chocolate, participants will undergo a similar sequence of exames after the consumption of white chocolate.

DETAILED DESCRIPTION:
Many studies have been carried out to investigate the possible effects of dark chocolate on our body.

Especially dark chocolate (DC) has been studied because it contains large quantities of cocoa and flavonoids. Regular cocoa consumption (dark chocolate) has antihypertensive and anti-inflammatory effects. A previous study demonstrated that dark chocolate may also have cardiovascular benefits. Their study showed that the consumption of DC (70% cocoa) induces vasodilation of the coronary arteries. In a cross-over study performed in 2013 by the PI of this study, dark chocolate (containing 70% cocoa) improved kidney oxygenation as assessed with renal MRI in healthy people two hours after its ingestion, whereas white chocolate did not induce any changes. The reasons for this increase remained hypothetical, as other aspects of renal physiology such as renal perfusion were not measured in this study. Chocolate intake also has potential side effects. As it is rich in calories and carbohydrates, long term, regular intake may lead to weight gain and its associated problems. Besides, the hemodynamic effects on DC intake in patients suffering from chronic kidney diseases (CKD) are also largely unknown. Hence, more insight in the renal physiological effects of DC intake is needed before any recommendation can be made on the potential usefulness of randomized controlled trials to test short-and long-term renal effects of DC intake.

Renal physiology, especially perfusion, can be monitored using renal ultrasound thanks to its Doppler mode. In particular, the renal resistive index (RRI) of intra-renal segmentary arteries is an interesting parameter in this context. RRI is defined as the difference between maximum systolic and minimum diastolic velocity divided by the maximum systolic velocity. RRI stands for the resistance that blood faces when passing through the kidneys. From a physiological viewpoint, vasoconstriction of intra-renal segmentary and interlobar arteries will increase RRI, whereas vasodilation of the main renal arteries will decrease the RRI. As chocolate induce vasodilatation of arteries, RRI is expected to decrease after DC intake.

Renal perfusion is also affected by the sympathetic nervous system, as its activation generates vasoconstriction of peripherical arteries, and possibly of the renal arteries. The handgrip test is a way to activate the sympathetic nervous system. With this test, volunteer applies an isometric strength with his hand to a handgrip device, which activates the sympathetic nervous system. . Therefore, the handgrip test can there be seen as a renal vascular stress test, but its effects on the RRI have not been studied. Besides, whether the RRI is influenced by the hand grip test, and whether this change is altered by DC intake, is also unknown. The handgrip test will therefore be used in the present study.

The aim of the present randomized controlled trial study is to investigate changes that may occur in kidneys after eating white and dark chocolate, as well as to see how renal perfusion works in this context and to evaluate responses to renal vascular stress (handgrip test). The innovation of the present study stands in the fact that the effect of chocolate intake on renal physiology has, to the best of our knowledge, not been investigated using renal ultrasound. It is also unknown whether the intake of chocolate may balance the renal physiology changes in response to stress (i.e. handgrip test).

ELIGIBILITY:
Inclusion Criteria for healthy volunteers:

* Age ≥ 18 years old
* ability to understand the study protocol and to sign an informed consent.

Inclusion criteria for CKD patients:

* Age ≥18 years old,
* CKD stage 1-3,
* ability to understand the study protocol and to sign an informed consent

Exclusion Criteria:

* Lactose or cocoa intolerance,
* Diabetes,
* any severe digestive issue and liver disease,
* history of kidney stones,
* inability to follow the procedures of the study, e.g. due to language problems, dementia, etc.
* pregnant women
* healthy volunteers taking antihypertensive medication
* healthy volunteers having a known kidney malformation or abnormality
* healthy volunteers with albuminuria and/or hematuria in the urine sample.
* CKD patients with an eGFR<30ml/min/1.73m2
* CKD patients with measured kalemia of > 5.5mmol/l in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Renal Resistive Index (RRI) | baseline versus 2 hours after DC or WC ingestion
  assess the differences in Doppler ultrasound- assessed RRI depending on the type of chocolate eaten by participants

SECONDARY OUTCOMES:
Peak Systolic Velocity (PSV) | baseline versus 2 hours after DC or WC ingestion
  assess the differences in Doppler-ultrasound assessed PSV depending on the type of chocolate eaten by participants
Peak Diastolic Velocity (PDV) | baseline versus 2 hours after DC or WC ingestion
  assess the differences in Doppler-ultrasound assessed PDV depending on the type of chocolate eaten by participants
Pulsatility Index (PuI) | baseline versus 2 hours after DC or WC ingestion
  assess the differences in Doppler-ultrasound assessed PuI depending on the type of chocolate eaten by participants
Systolic Blood Pressure (SBP) | baseline versus 2 hours after DC or WC ingestion
  assess the differences in Finapress-assessed SBP depending on the type of chocolate eaten by participants
Diastolic Blood Pressure (DBP) | baseline versus 2 hours after DC or WC ingestion
  assess the differences in Finapress-assessed DBP depending on the type of chocolate eaten by participants
Mean Arterial Pressure (MAP) | baseline versus 2 hours after DC or WC ingestion
  assess the differences in Finapress-assessed MAP depending on the type of chocolate eaten by participants
Handgrip-induced changes in RRI | baseline versus 2 hours after DC or WC ingestion
  assess the differences in handgrip-induced change in RRI depending on the type of chocolate eaten by participants

CONTACTS AND LOCATIONS:
Overall Officials: Menno Pruijm, PD MD, Principal Investigator — CHUV
Locations (2):
- Switzerland (2):
  - Department of Nephrology, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - University Hospital of Lausanne (CHUV), Lausanne, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grassi D, Necozione S, Lippi C, Croce G, Valeri L, Pasqualetti P, Desideri G, Blumberg JB, Ferri C. Cocoa reduces blood pressure and insulin resistance and improves endothelium-dependent vasodilation in hypertensives. Hypertension. 2005 Aug;46(2):398-405. doi: 10.1161/01.HYP.0000174990.46027.70. Epub 2005 Jul 18. PMID 16027246
- [Background] Fanton S, Cardozo LFMF, Combet E, Shiels PG, Stenvinkel P, Vieira IO, Narciso HR, Schmitz J, Mafra D. The sweet side of dark chocolate for chronic kidney disease patients. Clin Nutr. 2021 Jan;40(1):15-26. doi: 10.1016/j.clnu.2020.06.039. Epub 2020 Jul 14. PMID 32718711
- [Background] Flammer AJ, Hermann F, Sudano I, Spieker L, Hermann M, Cooper KA, Serafini M, Luscher TF, Ruschitzka F, Noll G, Corti R. Dark chocolate improves coronary vasomotion and reduces platelet reactivity. Circulation. 2007 Nov 20;116(21):2376-82. doi: 10.1161/CIRCULATIONAHA.107.713867. Epub 2007 Nov 5. PMID 17984375
- [Background] Buijsse B, Feskens EJ, Kok FJ, Kromhout D. Cocoa intake, blood pressure, and cardiovascular mortality: the Zutphen Elderly Study. Arch Intern Med. 2006 Feb 27;166(4):411-7. doi: 10.1001/archinte.166.4.411. PMID 16505260
- [Background] Pruijm M, Hofmann L, Charollais-Thoenig J, Forni V, Maillard M, Coristine A, Stuber M, Burnier M, Vogt B. Effect of dark chocolate on renal tissue oxygenation as measured by BOLD-MRI in healthy volunteers. Clin Nephrol. 2013 Sep;80(3):211-7. doi: 10.5414/CN107897. PMID 23557792